CLINICAL TRIAL: NCT01735760
Title: Comparison of Ultrasound Examination and Palpation to Locate the Cricothyroid Membrane - a Randomized Study
Brief Title: Ultrasound Examination Versus Palpation to Locate the Cricothyroid Membrane
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Seltz Kristensen, M.D., Rigshospitalet, Denmark
Other Study IDs: US-MC-001
Record Dates: First submitted 2012-11-24; First posted 2012-11-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Focus: Localizing the Cricothyroid Membrane Before Airway Management
Keywords: airway management; cricothyroid membrane

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Palpation: The group using palpation as primary attempt at localizing the cricothyroid membrane
- Ultrasonography: The group using ultrasound for their primary approach to localizing the cricothyroid membrane

SUMMARY:
Anesthesiologists get a course on localizing the cricothyroid membrane on a human using ultrasonography. Thereafter their ability to localize the cricothyroid membrane with either palpation or ultrasonography, in a randomised fashion, is tested.

DETAILED DESCRIPTION:
The ability to localize the cricothyroid membrane on patients before airway management is crucial in order to be able to follow the difficult airway algorithms.

Studies have show a high failure rate when anesthesiologists rely on palpation.

In this study Anesthesiologists get an e-learning course, get literature to study , and get a theoretical course and a hands-on course in using ultrasound for localizing the cricothyroid membrane. . Thereafter their ability to localize the cricothyroid membrane with either palpation or ultrasonography, in a randomised fashion, is tested.

ELIGIBILITY:
Inclusion Criteria:

* being an anesthesiologist attending our airway management course

Exclusion Criteria:

* unwillingness to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: anesthesiologists
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
rate of success of localizing the cricothyroid membrane with ultrasound and palpation | december 2012
  the rate of success is measured

SECONDARY OUTCOMES:
time to localise the cricothyroid membrane with ultrasonography and palpation | december 2012
  time measure for both ultrasonographic and palpation method

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Denmark, Copenhagen, Denmark